CLINICAL TRIAL: NCT00193596
Title: A Randomized, Phase III Comparison of Gemcitabine/Irinotecan Followed by IRESSA Versus Paclitaxel/Carboplatin/Etoposide Followed by IRESSA in the First-Line Treatment of Patients With Carcinoma of Unknown Primary Site
Brief Title: Gemcitabine/Irinotecan/ZD1839 vs Paclitaxel/Carboplatin/Etoposide/ZD1839 in Carcinoma of Unknown Primary Site
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: AstraZeneca (Industry); Pharmacia and Upjohn (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI UNKPRI 12
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: Neoplasms, Unknown Primary
Keywords: Neoplasms, Unknown Primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Etoposide; etoposide phosphate; Gemcitabine; Irinotecan; Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen A (Experimental): Paclitaxel 200 mg/m2 by 1-hour IV infusion, day 1
  Carboplatin area under the curve (AUC) 6.0 IV, day 1
  Etoposide 50 mg alternating with 100 mg by mouth, days 1 and 10
  Regimen A was repeated at a 21-day interval
  Interventions: Drug: Etoposide; Drug: Paclitaxel; Drug: Carboplatin
- Regimen B (Experimental): Irinotecan 100 mg/m2 IV, days 1 and 8
  Gemcitabine 1000 mg/m2 IV, days 1 and 8
  Regimen B was repeated at a 21-day interval
  Interventions: Drug: Gemcitabine; Drug: Irinotecan

INTERVENTIONS:
Drug: Etoposide — 50 mg alternating with 100 mg PO, days 1 and 10 in regimen A
  Other Names: Etopophos; Toposar
  Arms: Regimen A
Drug: Gemcitabine — 1000 mg/m2 IV, days 1 and 8, in regimen B
  Other Names: Gemzar
  Arms: Regimen B
Drug: Irinotecan — 1000 mg/m2 IV days 1 and 8 in regimen B
  Other Names: Camptosar
  Arms: Regimen B
Drug: Paclitaxel — 200 mg/m2 by 1-hour IV infusion, day 1, regimen A
  Other Names: Abraxane
  Arms: Regimen A
Drug: Carboplatin — Area under the curve (AUC) 6.0 IV, day 1, regimen A
  Other Names: Paraplatin
  Arms: Regimen A

SUMMARY:
In this randomized trial, we will investigate the activity and toxicity of two active regimens, gemcitabine/irinotecan and paclitaxel/carboplatin/Etoposide (both followed by ZD1839) in the first-line treatment of patients with carcinoma of unknown primary site.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be randomly assigned to one of two treatment arms:

* Paclitaxel + Carboplatin + Etoposide
* Irinotecan + Gemcitabine

Patients will be stratified by tumor location (liver/bone versus all others) and number of metastatic sites (one versus two or more). Patients with an objective response or stable disease after completion of chemotherapy will receive ZD1839 until disease progression. Patients who do not respond to chemotherapy may crossover to the other chemotherapy regimen and will receive ZD1839 if they have an objective response or stable disease. The study is not blinded so both the patient and the doctor will know which treatment has been assigned.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Carcinoma of unknown primary site
* Biopsy-proven metastatic carcinoma
* Able to perform activities of daily living with minimal assistance
* No previous treatment with any systemic therapy
* Measurable or evaluable disease
* Adequate bone marrow, liver and kidney function
* Understand the nature of this study and give written informed consent

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* Uncontrolled brain metastases and meningeal involvement
* Other uncontrolled malignancies
* Women pregnant or lactating
* Recent history of significant cardiovascular disease
* Severe or uncontrolled systemic disease
* Other significant clinical disorder
* Clinically active interstitial lung disease

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2003-09; Primary Completion 2008-09 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (31):
- United States (31):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Southern Cancer Center, Sacred Heart Heath System Medical Oncology Group, Mobile, Alabama
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Tower Oncology, Beverly Hills, California
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Mercy Hospital Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Phoebe Cancer Center, Albany, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Terrebonne General Medical Center, Houma, Louisiana
  - Mercy Hospital, Portland, Maine
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - St. Joseph Mercy Oakland Hospital, Cancer Center, Pontiac, Michigan
  - Jackson Oncology Associates, Jackson, Mississippi
  - Montana Cancer Institute Foundation, Missoula, Montana
  - Methodist Cancer Center, Omaha, Nebraska
  - Aultman Hospital, Canton, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Consultants in Medical Oncology and Hematology, Drexel Hill, Pennsylvania
  - Reading Hospital Regional Cancer Center, West Reading, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Kingsport Hematology-Oncology, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Cancer Outreach Associates, Abingdon, Virginia

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Clark BL, Shipley D, Thompson DS, Farley C, West-Osterfield K, Lane CM, Cescon T, Bury MJ, Greco FA. Paclitaxel/carboplatin/etoposide versus gemcitabine/irinotecan in the first-line treatment of patients with carcinoma of unknown primary site: a randomized, phase III Sarah Cannon Oncology Research Consortium Trial. Cancer J. 2010 Jan-Feb;16(1):70-5. doi: 10.1097/PPO.0b013e3181c6aa89. PMID 20164695
- See also: Published article in The Cancer Journal — http://journals.lww.com/journalppo/pages/articleviewer.aspx?year=2010&issue=02000&article=00013&type=abstract

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel/Carboplatin/Etoposide/Gefitinib: Paclitaxel 200 mg/m2 by 1-hour IV infusion, day 1
  Carboplatin area under the curve (AUC) 6.0 IV, day 1
  Etoposide 50 mg alternating with 100 mg by mouth, days 1 and 10
  Regimen A was repeated at a 21-day interval
- Irinotecan/Gemcitabine/Gefitinib: Irinotecan 100 mg/m2 IV, days 1 and 8
  Gemcitabine 1000 mg/m2 IV, days 1 and 8
  Regimen B was repeated at a 21-day interval
Period: Overall Study
Arm/Group | Paclitaxel/Carboplatin/Etoposide/Gefitinib | Irinotecan/Gemcitabine/Gefitinib
Started | 93 | 105
Completed | 37 | 39
Not Completed | 56 | 66

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel/Carboplatin/Etoposide/Gefitinib | Irinotecan/Gemcitabine/Gefitinib | Total
Number analyzed (Participants) | 93 | 105 | 198
Age Continuous [Median (Full Range); unit: years] | 61 [39 to 82] | 59 [33 to 83] | 60 [33 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 42 | 91
  Male | 44 | 63 | 107
Region of Enrollment [Number; unit: participants]
  United States | 93 | 105 | 198

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Description: Length of time, in months, that patients were alive from their first date of protocol treatment until death.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/Carboplatin/Etoposide/Gefitinib | Irinotecan/Gemcitabine/Gefitinib
Number analyzed (Participants) | 93 | 105
months | 7.4 [4.67 to 10.28] | 8.5 [6.64 to 10.58]

2. Secondary Outcome: Progression Free Survival (PFS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease
Description: Length of time, in months, that patients were alive from their first date of protocol treatment until worsening of their disease
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/Carboplatin/Etoposide/Gefitinib | Irinotecan/Gemcitabine/Gefitinib
Number analyzed (Participants) | 93 | 105
months | 3.3 [2.2 to 4.86] | 5.3 [3.88 to 6.21]

ADVERSE EVENTS:
Arm/Group | Paclitaxel/Carboplatin/Etoposide/Gefitinib | Irinotecan/Gemcitabine/Gefitinib
Serious Adverse Events (participants affected / at risk) | 56/93 | 57/105
Other Adverse Events (participants affected / at risk) | 93/93 | 105/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel/Carboplatin/Etoposide/Gefitinib (N=93) | Irinotecan/Gemcitabine/Gefitinib (N=105)
Ocular - Other (Eye disorders) | 1 (1) | 0 (0) — Temporary unilateral blindness
Febrile Neutropenia (Infections and infestations) | 16 (16) | 5 (5)
Death (General disorders) | 9 (9) | 8 (8)
Infection - Skin (Infections and infestations) | 1 (1) | 2 (2)
Infection - Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Superventricular Arrhythmia - Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Pain - Abdomen (General disorders) | 1 (1) | 3 (3)
Dehydration (Gastrointestinal disorders) | 7 (8) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infection with Unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 (2) | 5 (5)
Infection - GI (Infections and infestations) | 0 (0) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 2 (2) | 3 (3)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neurology - Other (Nervous system disorders) | 1 (1) | 0 (0) — Cauda Equina Syndrome
Pulmonary - COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 4 (5)
Spinal Cord Compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Confusion (Nervous system disorders) | 2 (3) | 2 (2)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Pulmonary - Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstruction - Bile Duct (Hepatobiliary disorders) | 2 (2) | 1 (1)
Respiratary - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Interstitial lung changes
Ulcer, GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infection - Renal/Genitourinary (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Obstruction - GI (Gastrointestinal disorders) | 0 (0) | 2 (2)
Infection - Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
GI - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) — Ischemic Bowel
Edema: Head and Neck (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (2)
Valvular Heart Disease (Cardiac disorders) | 1 (1) | 0 (0)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Peripheal Arterial Ischemia (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vasovagal Episode (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver Dysfunction (Hepatobiliary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel/Carboplatin/Etoposide/Gefitinib (N=93) | Irinotecan/Gemcitabine/Gefitinib (N=105)
Alopecia (Skin and subcutaneous tissue disorders) | 70 (243) | 45 (130)
Anorexia (Gastrointestinal disorders) | 58 (108) | 66 (141)
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 (80) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 36 (65)
Diarrhea (Gastrointestinal disorders) | 42 (67) | 61 (115)
Edema - NOS (Blood and lymphatic system disorders) | 25 (44) | 34 (74)
Fatigue (General disorders) | 93 (300) | 105 (363)
Febrile Neutropenia (Infections and infestations) | 30 (32) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 58 (138) | 60 (137)
Infection - NOS (Infections and infestations) | 29 (38) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 55 (160) | 51 (143)
Mucositis/Stomatitis (Gastrointestinal disorders) | 25 (39) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 27 (46) | 0 (0)
Nausea (Gastrointestinal disorders) | 82 (164) | 85 (196)
Neuropathy (Nervous system disorders) | 50 (143) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 52 (115) | 32 (84)
Pain (General disorders) | 71 (164) | 80 (163)
Pulmonary - NOS (Respiratory, thoracic and mediastinal disorders) | 39 (67) | 40 (82)
Vomiting (Gastrointestinal disorders) | 48 (70) | 48 (79)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.